CLINICAL TRIAL: NCT05444465
Title: Evaluation of Safety and Efficacy of a Resorbable Collagen Implant in Treatment of High Grade PArtial ThiCkness Tears; A Prospective, Multicenter, Randomized, Control Trial (IMPACT Study)
Brief Title: Use of the REGENETEN™ Bioinductive Implant System in High Grade Partial-thickness Tears
Acronym: IMPACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REGENETEN.2021.04
Record Dates: First submitted 2022-06-29; First posted 2022-07-06 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Rotator Cuff Injuries
Keywords: Rotator cuff tear; High grade partial thickness tears; REGENETEN Bioinductive Implant System
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Wound Healing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Isolated Bioinductive Repair (Experimental): Surgical treatment of partial-thickness rotator cuff tears with the REGENETEN Bioinductive Implant system.
  Interventions: Device: Isolated Bioinductive Repair
- Completion and Repair (Active Comparator): Surgical treatment of partial-thickness rotator cuff tears using the standard surgical technique 'Completion and Repair'.
  Interventions: Procedure: Completion and Repair

INTERVENTIONS:
Device: Isolated Bioinductive Repair — Isolated Bioinductive repair with REGENETEN™ Bioinductive Implant
  Other Names: REGENETEN™ Bioinductive Implant
  Arms: Isolated Bioinductive Repair
Procedure: Completion and Repair — Standard surgical repair using the 'Completion and Repair' technique.
  Arms: Completion and Repair

SUMMARY:
The purpose of the study is to assess whether the REGENETEN™ Bioinductive Implant allows patients to get back to their everyday activities quicker than if the tendon is repaired by the standard repair technique 'Completion and Repair' for surgically treating partial-thickness rotator cuff tears.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the functional recovery of patients with high grade (>50%) partial thickness tears at 3 months when treated with either Isolated Bioinductive Repair (IBR) or Completion and Repair (CAR).

ELIGIBILITY:
Inclusion Criteria:

* The subject must provide written informed consent.
* Subject is > eighteen (18) years of age (no upper limit).
* Subject has an isolated high-grade (>50% or >6mm) (Ellman grade III) partial thickness tear of supraspinatus or supraspinatus with infraspinatus.
* Subject has failed a minimum of 3 months of conservative management for treatment of partial thickness rotator cuff tear.
* Subject willing and able to make all required study visits.
* Subject able to follow instructions and deemed capable of completing all study questionnaires.

Exclusion Criteria:

* Subjects with insufficient tendon tissue quality for management and protection of the tendon injury using the isolated REGENETEN Bioinductive Implant system.
* Subjects where the prescribed Physical Therapy guidelines stated in the protocol are not suitable for their rehabilitation.
* Subjects with Samilson-Prieto osteoarthritis grade 2 and greater.
* Subjects with current or prior infection of the ipsilateral shoulder.
* Subjects with known hypersensitivity to bovine-derived materials.
* Subjects with known inflammatory arthropathy, history of inflammatory arthropathy, chronic joint disease or chronic pain of upper extremities (shoulder(s), arm(s)).
* Subjects with prior shoulder surgery on index shoulder, including subacromial decompression, biceps tenodesis/tenotomy, and acromioclavicular joint (ACJ) excision/distal clavicle excision (DCE).
* Subjects with a planned surgery on the contra-lateral shoulder within the study period.
* Systemic steroid use (oral, IV) or local steroid injection within 3 months of the date of surgery.
* Subjects with a full thickness rotator cuff tear.
* Subjects with a subscapularis tear requiring repair.
* Subjects requiring a concomitant labral fixation procedure, concomitant surgery for bone defects requiring bone implantation or for superior labral tear from anterior to posterior (SLAP).
* Subjects requiring a concomitant os acromiale fixation procedure.
* Subjects with glenohumeral joint instability (multiple dislocations/subluxations).
* Subjects with condition(s) that contraindicate or complicate outcomes of Isolated Bioinductive Repair or completion and repair e.g., > Hamada 3 rotator cuff arthropathy on X-ray, Goutallier atrophy > Grade 3, proximal humeral fracture or scapular fracture, avascular necrosis of the humeral head.
* Subjects with neurologic conditions effecting either upper extremity.
* Subjects who are unable to tolerate magnetic resonance imaging (MRI), due to psychiatric or medical contraindications.
* Subjects who are pregnant or breast feeding.
* Subjects who are currently involved in any injury litigation relating to the index shoulder.
* Subjects with current workers compensation claim.
* Subjects who are enrolled, or plan to enroll, in another clinical trial during this study that would affect the outcomes of this study.
* Subjects with a history of poor compliance with medical treatment, physical therapy (PT)/rehabilitation, or clinical study participation.
* Subject who, in the opinion of the Investigator, has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, mental retardation, and drug or alcohol abuse.
* Subjects who do not meet the indication or are contraindicated according to specific Smith+Nephew REGENETEN System's Instructions for Use (IFUs).
* Any subject that meets the definition of a Vulnerable Subject per ISO 14155 Section 3.55.
* Subjects who have participated previously in this clinical trial and who have healed or been withdrawn
* Subjects with a medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Western Ontario Rotator Cuff (WORC) | Change from baseline to 3 months post-intervention
  The WORC Index is self-administered, and includes a 5 different domains (physical symptoms, sports and recreation, work, social function, and emotions). Each question uses a visual analog scale (VAS) representing a 100-point scale ranging from 0 to 100. The maximum score is 2100 (worst possible symptoms). Zero (0) represents no symptoms at all. The final score can also be presented as a percentage by subtracting the total from 2100, dividing by 2100, and multiplying by 100. This will give you an overall percentage. The total final WORC Index scores can, therefore, range from 0% (lowest functional status level) to 100% (highest functional status level).

SECONDARY OUTCOMES:
Western Ontario Rotator Cuff (WORC) | Pre-op, 6 weeks, 3, 6, 12 and 24 months
  The WORC Index is self-administered, and includes a 5 different domains (physical symptoms, sports and recreation, work, social function, and emotions). Each question uses a visual analog scale (VAS) representing a 100-point scale ranging from 0 to 100. The maximum score is 2100 (worst possible symptoms). Zero (0) represents no symptoms at all. The final score can also be presented as a percentage by subtracting the total from 2100, dividing by 2100, and multiplying by 100. This will give you an overall percentage. The total final WORC Index scores can, therefore, range from 0% (lowest functional status level) to 100% (highest functional status level).
Constant-Murley Score | Pre-Op, 3, 6, 12 and 24 months
  The Constant-Murley Score is a validated assessment of pain and shoulder functionality. The Constant Score is divided into 4 subscales: pain (15 points; VAS score range of 0-15), activities of daily living (20 points; range 0=worst, 5=best), strength (25 points; 1 point given per 0.5 kg of weights raised), and range of motion - forward flexion, external rotation, abduction and internal rotation of the shoulder (40 points; range 0=worst, 10=best). The higher the score, the higher the quality of function.
Subjective Shoulder Value (SSV) score | Pre-Op, 6 weeks, 3, 12 and 24 months
  The SSV is defined as a patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder, which would score 100% (0% to 100% scale with 100% being normal).
EuroQol 5 Dimension 5 Level (EQ-5D-5L) VAS & index scores | Pre-Op, 3 and 6 weeks, 3, 6, 12 and 24 months
  To assess the subject's health state. The EQ-5D-5L is composed of the EQ- 5D-5L descriptive system and the EQ Visual Analogue scale (EQ VAS).
  The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Responses are coded as single-digit numbers expressing the severity level selected in each dimension. For instance, 'slight problems' (e.g. 'I have slight problems in walking about') is always coded as '2'. The digits for the five dimensions are combined in a 5-digit code. The EQ- 5D-5L index value is derived by using the vendor supplied calculator to convert each 5-digit EQ- 5D-5L profile.
  The EQ VAS corresponds to a 20 cm vertical, visual analogue scale ranging from 'the best health you can imagine' to 'the worst health you can imagine'.
  A higher number is a better outcome.
Change in Western Ontario Rotator Cuff (WORC) | Change from Pre-op to 6 weeks, 3, 6, 12 and 24 months
  The WORC Index is self-administered, and includes a 5 different domains (physical symptoms, sports and recreation, work, social function, and emotions). Each question uses a visual analog scale (VAS) representing a 100-point scale ranging from 0 to 100. The maximum score is 2100 (worst possible symptoms). Zero (0) represents no symptoms at all. The final score can also be presented as a percentage by subtracting the total from 2100, dividing by 2100, and multiplying by 100. This will give you an overall percentage. The total final WORC Index scores can, therefore, range from 0% (lowest functional status level) to 100% (highest functional status level).
Change in Constant-Murley Score | Change from Pre-Op to 6 weeks, 3, 12 and 24 months
  The Constant-Murley Score is a validated assessment of pain and shoulder functionality. The Constant Score is divided into 4 subscales: pain (15 points; VAS score range of 0-15), activities of daily living (20 points; range 0=worst, 5=best), strength (25 points; 1 point given per 0.5 kg of weights raised), and range of motion - forward flexion, external rotation, abduction and internal rotation of the shoulder (40 points; range 0=worst, 10=best). The higher the score, the higher the quality of function.
Change in Subjective Shoulder Value (SSV) score | Change from Pre-Op to 6 weeks, 3, 12 and 24 months
  The SSV is defined as a patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder, which would score 100% (0% to 100% scale with 100% being normal).
Percent Achieving Minimal Clinically Important Difference (MCID) for Constant-Murley Score | Pre-Op, 3, 6, 12 and 24 months
  The Constant-Murley Score is a validated assessment of pain and shoulder functionality. The Constant Score is divided into 4 subscales: pain (15 points; VAS score range of 0-15), activities of daily living (20 points; range 0=worst, 5=best), strength (25 points; 1 point given per 0.5 kg of weights raised), and range of motion - forward flexion, external rotation, abduction and internal rotation of the shoulder (40 points; range 0=worst, 10=best). The higher the score, the higher the quality of function.
Percent Achieving MCID for Western Ontario Rotator Cuff (WORC) | Pre-op, 6 weeks, 3, 6, 12 and 24 months
  The WORC Index is self-administered, and includes a 5 different domains (physical symptoms, sports and recreation, work, social function, and emotions). Each question uses a visual analog scale (VAS) representing a 100-point scale ranging from 0 to 100. The maximum score is 2100 (worst possible symptoms). Zero (0) represents no symptoms at all. The final score can also be presented as a percentage by subtracting the total from 2100, dividing by 2100, and multiplying by 100. This will give you an overall percentage. The total final WORC Index scores can, therefore, range from 0% (lowest functional status level) to 100% (highest functional status level).
Percent Achieving MCID for Subjective Shoulder Value (SSV) score | Pre-Op, 6 weeks, 3, 12 and 24 months
  The SSV is defined as a patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder, which would score 100% (0% to 100% scale with 100% being normal).
Patient Satisfaction | 6 weeks, 3, 6, 12 and 24 months
  Comprise of 2 questions:
  1. Overall, I am satisfied with the outcome of my surgery
  2. I would recommend the procedure to a friend.
  Question rated by the patient with Strongly Agree, Agree, Neither Agree nor Disagree, Disagree, Strongly Disagree.
Pain, Visual analog scale (VAS) Score | Pre-Op, 3 and 6 weeks, 3, 12 and 24 months
  Pain is assessed on a 100-point scale ranging from 0 to 100, with zero (0) representing no pain and 100 representing the worst pain imaginable.
MRI Tendon Findings in subjects with Isolated Bioinductive Repair versus completion via Sugaya Score | 12 months
  The Sugaya score is classified into 5 categories: Type I to Type V. Type I indicates sufficient thickness with homogenously low intensity. Type II indicates sufficient thickness with partial high intensity. Type III indicates insufficient thickness without discontinuity. Type IV indicates presence of a minor discontinuity, suggesting a small full-thickness tear. Type V indicates the presence of a major discontinuity, suggesting a medium or large full-thickness tear.
MRI Tendon Findings in subjects with Isolated Bioinductive Repair versus completion via MRI assessment of percent filling | 12 months
  Percent tissue infil is graded at site of original tear and classified as 0% to < 25%, 25% to < 50%, 50% to < 75%, 75% to < 100% and 100%.
MRI Tendon Findings in subjects with Isolated Bioinductive Repair versus completion via MRI assessment of the signal intensity pattern | 12 months
  The Signal Intensity Pattern will be graded into 3 categories. Type I: Heterogeneous high signal intensity with fluid-like bright foci, Type II: Heterogeneous high signal intensity without fluid-like bright foci, Type III: Heterogeneous or homogeneous low signal intensity.
MRI Tendon Findings in subjects with Isolated Bioinductive Repair versus completion via Rotator cuff tendon thickness | 12 months
  Tendon thickness will be measured in millimeters (mm).
MRI Tendon Findings in subjects with Isolated Bioinductive Repair versus completion via Goutallier classification | 12 months
  The Goutallier classification will be used to classify the fatty infiltration of the rotator cuff. The Goutallier classification ranges from a grade of 0 indicating a completely normal muscles without any fatty streaks to a grade of 4 which indicates that more fat than muscle is present.
Incidence of Revision Surgery | 1, 3 and 6 weeks, 3, 6, 12 and 24 months
  Number of subjects requiring revision surgery
Time to return to work | Up to 24 months
  Number of weeks taken to return to work following surgery
Time to return to driving | Up to 24 months
  Number of weeks taken to return to driving following surgery
Time to return to sports | Up to 24 months
  Number of weeks taken to return to sport following surgery
Total operative time | Inter-operative time
  Time expressed in minutes
Physical Therapy Utilization | Up to 24 months
  Number visits following index surgery
Cumulative days of opioid use | Day 1-14
  Self-reported opioid use diary completed by the patient on a daily basis, from day 0-14, documenting opioid use. Consumption daily (YES/NO) x14 days, 'Have you taken any opioid medication today for shoulder pain?'
Duration of shoulder immobilization following index surgery | 1, 3 and 6 weeks, 3 months
  Number of days

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mills, Study Chair — Smith & Nephew, Inc.
Locations (20):
- United States (8):
  - Harbin Clinic, Rome, Georgia
  - OrthoIllinois LTD, Rockford, Illinois
  - Sinai Hospital Baltimore, Baltimore, Maryland
  - Cleveland Clinic - Sports Health, Garfield Heights, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Orthopedic Specialists, Bedford, Texas
  - Houston Methodist The Woodlands, The Woodlands, Texas
  - Memorial Medical Center, Ashland, Wisconsin
- OrthoSport Victoria, Richmond, Victoria, Australia
- Canada (3):
  - Access Orthopaedics, Calgary, Alberta
  - Pan Am Clinic, Winnipeg, Manitoba
  - Research St. Joseph's, Hamilton, Ontario
- Italy (2):
  - IRCCS Istituto Ortopedico Galeazzi,, Milan
  - Fondazione Policlinico Universitario Campus Bio-Medico, Roma
- Spain (2):
  - Hospital Ramón y Cajal, Madrid
  - Hospital Fundación Jiménez Díaz, Madrid
- United Kingdom (4):
  - Ashford & St Peter's Hospitals NHS Foundation Trust, Chertsey, Surrey
  - Sulis Hospital, Bath
  - North Bristol NHS Trust, Bristol
  - Northern Care Alliance NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: No